CLINICAL TRIAL: NCT01173874
Title: Clinical and Biomarker Assessment of Efficacy of Cognitive Remediation in Patients With Schizophrenia or Schizoaffective Disorder Stabilized on Lurasidone
Brief Title: Efficacy of Cognitive Remediation in Patients With Schizophrenia or Schizoaffective Disorder Stabilized on Lurasidone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #6121
Record Dates: First submitted 2010-07-08; First posted 2010-08-02 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Schizophrenia
Keywords: Cognition; Function; Attention; Vigilance; Verbal Memory; Visual Memory; Processing Speed; Problem Solving; Social Cognition
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Remediation (Experimental): Cognitive remediation intervention will be administered in small group settings twice weekly for 30 sessions and will utilize computerized and verbal group training exercises to address basic skills such as auditory processing, attention, processing speed, and verbal working memory and learning, as well as intermediate and complex skills such as deductive reasoning, planning and sequencing, set shifting, and complex problem solving.
  Interventions: Drug: Cognitive Remediation
- Cognitive activity control group (No Intervention): This is a non-specific mental activity control condition, conducted two times per week for a total of 30 sessions.

INTERVENTIONS:
Drug: Cognitive Remediation — Cognitive remediation intervention will be administered in small group settings twice weekly for 30 sessions and will utilize computerized and verbal group training exercises to address basic skills such as auditory processing, attention, processing speed, and verbal working memory and learning, as well as intermediate and complex skills such as deductive reasoning, planning and sequencing, set shifting, and complex problem solving.
  Arms: Cognitive Remediation

SUMMARY:
The investigators hypothesize that cognitive remediation will be superior to the active control group on the change from baseline to study end point of cognitive remediation phase on both co-primary outcome measures (standardized composite MATRICS score and Cognitive Assessment Interview).

DETAILED DESCRIPTION:
OVERVIEW & SPECIFIC AIMS Marked cognitive impairment underlies much of the social & occupational dysfunction associated with schizophrenia. Currently available antipsychotic medications are primarily effective in treating psychotic symptoms & have demonstrated only limited potential in ameliorating cognitive deficits in schizophrenia patients.

Lurasidone is a novel compound synthesized by SEPRACOR, Inc.for the treatment of patients with schizophrenia & bipolar disorder. It possesses high affinity for dopamine D2, serotonin 5-HT2A, 5-HT7, 5-HT1A & noradrenaline α2C receptors. Compared with other atypical antipsychotics, lurasidone demonstrates similar binding affinities for the D2 & 5-HT2A receptors, but greater affinity for serotonin 5-HT1A receptors. Lurasidone displays no affinity for histamine H1 or acetylcholine M1 receptors. In animal studies, lurasidone significantly reversed memory impairment induced by MK-801, an N-methyl-D-aspartate (NMDA) receptor antagonist, in a rat step-through type passive avoidance task. The maximum inhibitory effects of lurasidone were greater than those observed with risperidone, quetiapine, & olanzapine, while aripiprazole was not effective in reversing the impairment induced by MK-801. Additionally, lurasidone significantly reversed memory impairment induced by the anticholinergic drug scopolamine in the passive avoidance task. The reversal of pharmacologically induced cognitive deficits in rats by lurasidone is promising & warrants specific investigation in subjects with schizophrenia, given the prominence of cognitive deficits in this disorder.

From a different therapeutic perspective, the utility of cognitive remediation in ameliorating cognitive deficits & improving functional outcomes in schizophrenia has recently been evaluated in several studies. A meta-analysis of these trials found effect sizes for improvement in cognitive & psychosocial functioning in the low to moderate range (McGurck 2007). The best outcomes in psychosocial functioning were evident when cognitive remediation was combined with teaching of psychosocial skills.

Given the recalcitrant nature of cognitive deficits in schizophrenia & their impact on functional capacity we felt that in designing a study to test the effectiveness of cognitive remediation we should maximize the likelihood of therapeutic benefit by administering cognitive remediation in the context of pharmacotherapy that may have potential for precognitive effects. By so doing we could possibly boost the effect sizes seen with cognitive remediation alone. In this study we will transition patients with schizophrenia (in whom a change in antipsychotic therapy is clinically warranted) from their current antipsychotic to lurasidone - clinicians will have eight weeks to complete the switch. Subjects who are successfully switched to lurasidone will then be randomized to receive either cognitive remediation or a non-specific mental activity control condition two times/week for a total of 30 sessions over a 4-6 month period. Our goal is to have 140 patients complete the cognitive remediation phase.

A subset of the sample will participate in 2 biomarker studies. Event related potentials & fMRI will be done in these subjects at baseline & study completion.

This study will be done as an Investigator initiated trial (J. Lieberman, M.D. - PI) under a separate IND.

Primary Aim: We hypothesize that cognitive remediation will be superior to the active control group on the change from baseline to study end point of cognitive remediation phase on both co-primary outcome measures (standardized composite MATRICS score & Cognitive Assessment Interview).

Additional aims

1. To compare cognitive remediation to active control on functional outcome as assessed by the change in UCSD Performance-Based Skills Assessment (UPSA-Brief) from baseline to end point of cognitive remediation phase.
2. To compare cognitive remediation to active control on changes from lurasidone stabilized baseline to end point in indices of functional brain activation (ERP & fMRI) during cognitive activation tasks.
3. Evaluate the effect of 8 weeks of lurasidone treatment on cognitive & functional outcomes as assessed by changes from baseline in the MATRICS composite score, CAI, & UPSA-Brief.
4. Evaluate the effect of cognitive remediation compared to nonspecific mental activity on cognitive & functional outcomes as assessed by changes from lurasidone stabilized baseline to end of cognitive remediation phase in the MATRICS composite score, CAI, & UPSA-Brief.
5. Evaluate the efficacy, safety, & tolerability of lurasidone in patients with schizophrenia as assessed by the change from baseline to week 8 & to end of cognitive remediation phase in the PANSS total score, Side Effect Checklist, AIMS, SAS, BAS, & frequency of abnormal laboratory values.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18-55 years of age who meet DSM-IV-TR criteria for schizophrenia or schizoaffective disorder confirmed by the Structured Clinical Interview for DSM-IV Clinical trial version (SCID-CT version). Duration of illness > 1 year. Outpatient status.
* Change in antipsychotic medication is clinically warranted as evidenced by

  * persistent psychosis despite adequate dose and duration of antipsychotic, or * inability to achieve therapeutic dose because of dose-limiting side effects,
  * persistent side effects that either cause significant subjective distress or significantly increase medical risks, such as substantial weight gain or metabolic disturbances, or
  * patient preference to switch and treating psychiatrist is in agreement.
* No behaviors suggesting potential danger to self or others over the 6 months prior to participation.
* For the last 2 weeks of lurasidone stabilization phase, a score of 4 or less on PANSS items of conceptual disorganization, hallucinations, suspiciousness and unusual thought content items.
* At end of lurasidone stabilization phase, Simpson-Angus Scale total score <
* At end of lurasidone stabilization phase, Calgary Depression Scale total score <10.
* No acute medical problems; any chronic medical condition (e.g. hypertension) consistently treated and stable during the 1 month prior to participation.
* Able to provide signed informed consent and to cooperate with all study procedures.
* Able to attend twice weekly sessions (each lasting approximately 75 minutes) for cognitive remediation or active control sessions for the ~6 month duration of the cognitive remediation phase of the study.
* Must meet the following cognitive performance criteria:

  * Able to complete the baseline MATRICS validly at baseline as assessed by NP tester.
  * Raw score of 12 or greater on the WTAR (Wechsler Test of Adult Reading) at screening.
* Women who can become pregnant must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the study in such a manner that the risk of pregnancy is minimized. Acceptable methods include oral, injectable or implanted contraceptives, intrauterine devices or barrier methods such as condoms, diaphragm and spermicides. Women who can become pregnant must have a negative urine pregnancy test at the Screening Visit. Women who can become pregnant include anyone who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy), or is not postmenopausal (defined as amenorrhea 12 consecutive months).

Exclusion Criteria:

* Documented history of learning disability.
* Hearing or visual impairment; not fluent in English.
* Current treatment with clozapine or history of treatment resistance as evidenced by failure to improve (in the judgment of the investigator) with 2 or more adequate dose antipsychotic trials of at least 6 weeks duration in preceding 1 year.
* Concomitant or anticipated treatment with potent CYP 3A4 inhibitor such a cimetidine, cyclosporine, erythromycin or erythromycin-like drugs (e.g., azithromycin, clarithromycin except short term acute treatment for 1 week or less), diltiazem, itraconazole, ketoconazole or other systemic antifungal agents in the azole class, nefazodone; or potent CYP3A4 inducer including: carbamazepine, modafinil, Phenobarbital, phenytoin, rifampin, St. Johns Wort, and troglitazone.
* Current treatment with psychotropic agents known to affect cognition such as amphetamines, topiramate.
* History of treatment with electroconvulsive therapy within the 6 months prior to participation or expectation that patient may require ECT during the study.
* History of neurological or neuropsychiatric conditions (e.g. stroke, traumatic brain injury, epilepsy, etc).
* Subjects with a history of clinically significant neurological, metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, and/or urological disorders (e.g. unstable angina, decompensate congestive heart failure, CNS infection or history of HIV seropositivity), which would pose a risk to the patient if they were to participate in the study or that might confound the results of the study. Active medical conditions that are minor or well controlled are not exclusionary if they do not affect risk to the patient of the study results. For example, the following are not exclusionary: a) stable and well-controlled hypertension; b) asthma (no serious attacks in the past year); c) hypothyroidism (TSH within normal limits).
* A positive test for Hepatitis C antibody with concurrent evidence of impaired hepatic function (increased AST or ALT greater than 2 times the upper limit of normal) or positive tests for Hepatitis A antibody IgM fraction or Hepatitis B surface antigen, irrespective of the AST or ALT values.
* History of alcohol or substance abuse or dependence during the 6 months prior to participation.
* Participation in a clinical trial involving an investigational medication within 3 months prior to participation or 2 or more investigational drug trials in the preceding 12 months.
* Pregnant women or women of child-bearing potential who are not using adequate birth control.
* Woman who are breast feeding.
* Individuals who: a) received any cognitive remediation in the 6 months prior to study entry or b)received more than 6 hours of cognitive remediation in the 12 months prior to study entry or c) received more than 15 hours in the 24 months prior to study entry. Cognitive remediation is defined as any behavioral intervention consisting of training activities that aim to target impairments in cognitive domains of sensory processing, attention, memory, processing speed, working memory, and executive functioning.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-07; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lieberman, M.D., Principal Investigator — Columbia University; Zafar Sharif, M.D., Principal Investigator — Columbia University
Locations (16):
- United States (16):
  - San Fernando Mental Health Center, Granada Hills, California
  - University of California - Irvine, Orange, California
  - Yale University, New Haven, Connecticut
  - University of Miami Department of Psychiatry, Miami, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Psychiatric Clinical Research Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri, Columbia, Missouri
  - Columbia University, New York, New York
  - Psychopharmacology Research Unit- Nathan KIine Institute for Psychiatric Research, New York, New York
  - Duke University Medical Center, Butner, North Carolina
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center, San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baddeley A. Working memory. Science. 1992 Jan 31;255(5044):556-9. doi: 10.1126/science.1736359.
- [Background] Bruder GE, Wexler BE, Sage MM, Gil RB, Gorman JM. Verbal memory in schizophrenia: additional evidence of subtypes having different cognitive deficits. Schizophr Res. 2004 Jun 1;68(2-3):137-47. doi: 10.1016/S0920-9964(03)00156-7. PMID 15099598
- [Background] Carter CS, Perlstein W, Ganguli R, Brar J, Mintun M, Cohen JD. Functional hypofrontality and working memory dysfunction in schizophrenia. Am J Psychiatry. 1998 Sep;155(9):1285-7. doi: 10.1176/ajp.155.9.1285. PMID 9734557
- [Background] Davidson M, Galderisi S, Weiser M, Werbeloff N, Fleischhacker WW, Keefe RS, Boter H, Keet IP, Prelipceanu D, Rybakowski JK, Libiger J, Hummer M, Dollfus S, Lopez-Ibor JJ, Hranov LG, Gaebel W, Peuskens J, Lindefors N, Riecher-Rossler A, Kahn RS. Cognitive effects of antipsychotic drugs in first-episode schizophrenia and schizophreniform disorder: a randomized, open-label clinical trial (EUFEST). Am J Psychiatry. 2009 Jun;166(6):675-82. doi: 10.1176/appi.ajp.2008.08060806. Epub 2009 Apr 15. PMID 19369319
- [Background] Elger CE, Grunwald T, Lehnertz K, Kutas M, Helmstaedter C, Brockhaus A, Van Roost D, Heinze HJ. Human temporal lobe potentials in verbal learning and memory processes. Neuropsychologia. 1997 May;35(5):657-67. doi: 10.1016/s0028-3932(96)00110-8. PMID 9153028
- [Background] Fisher M, Holland C, Merzenich MM, Vinogradov S. Using neuroplasticity-based auditory training to improve verbal memory in schizophrenia. Am J Psychiatry. 2009 Jul;166(7):805-11. doi: 10.1176/appi.ajp.2009.08050757. Epub 2009 May 15. PMID 19448187
- [Background] Goldman-Rakic PS. The physiological approach: functional architecture of working memory and disordered cognition in schizophrenia. Biol Psychiatry. 1999 Sep 1;46(5):650-61. doi: 10.1016/s0006-3223(99)00130-4. PMID 10472417
- [Background] Goldman-Rakic PS. Working memory dysfunction in schizophrenia. J Neuropsychiatry Clin Neurosci. 1994 Fall;6(4):348-57. doi: 10.1176/jnp.6.4.348. PMID 7841806
- [Background] Green MF, Kern RS, Heaton RK. Longitudinal studies of cognition and functional outcome in schizophrenia: implications for MATRICS. Schizophr Res. 2004 Dec 15;72(1):41-51. doi: 10.1016/j.schres.2004.09.009. PMID 15531406
- [Background] Green MF. What are the functional consequences of neurocognitive deficits in schizophrenia? Am J Psychiatry. 1996 Mar;153(3):321-30. doi: 10.1176/ajp.153.3.321. PMID 8610818
- [Background] Gur RE, Jaggi JL, Shtasel DL, Ragland JD, Gur RC. Cerebral blood flow in schizophrenia: effects of memory processing on regional activation. Biol Psychiatry. 1994 Jan 1;35(1):3-15. doi: 10.1016/0006-3223(94)91160-6. PMID 8167200
- [Background] Kayser J, Bruder GE, Friedman D, Tenke CE, Amador XF, Clark SC, Malaspina D, Gorman JM. Brain event-related potentials (ERPs) in schizophrenia during a word recognition memory task. Int J Psychophysiol. 1999 Dec;34(3):249-65. doi: 10.1016/s0167-8760(99)00082-3. PMID 10610049
- [Background] Kayser J, Tenke CE. Principal components analysis of Laplacian waveforms as a generic method for identifying ERP generator patterns: I. Evaluation with auditory oddball tasks. Clin Neurophysiol. 2006 Feb;117(2):348-68. doi: 10.1016/j.clinph.2005.08.034. Epub 2005 Dec 13. PMID 16356767
- [Background] Kayser J, Tenke CE. Principal components analysis of Laplacian waveforms as a generic method for identifying ERP generator patterns: II. Adequacy of low-density estimates. Clin Neurophysiol. 2006 Feb;117(2):369-80. doi: 10.1016/j.clinph.2005.08.033. Epub 2005 Dec 13. PMID 16356768
- [Background] Kayser J, Tenke CE, Gates NA, Kroppmann CJ, Gil RB, Bruder GE. ERP/CSD indices of impaired verbal working memory subprocesses in schizophrenia. Psychophysiology. 2006 May;43(3):237-52. doi: 10.1111/j.1469-8986.2006.00398.x. PMID 16805862
- [Background] Kayser J, Tenke CE, Gates NA, Bruder GE. Reference-independent ERP old/new effects of auditory and visual word recognition memory: Joint extraction of stimulus- and response-locked neuronal generator patterns. Psychophysiology. 2007 Nov;44(6):949-67. doi: 10.1111/j.1469-8986.2007.00562.x. Epub 2007 Jul 19. PMID 17640266
- [Background] Sambataro F, Reed JD, Murty VP, Das S, Tan HY, Callicott JH, Weinberger DR, Mattay VS. Catechol-O-methyltransferase valine(158)methionine polymorphism modulates brain networks underlying working memory across adulthood. Biol Psychiatry. 2009 Sep 15;66(6):540-8. doi: 10.1016/j.biopsych.2009.04.014. Epub 2009 Jun 17. PMID 19539269
- [Background] McGurk SR, Twamley EW, Sitzer DI, McHugo GJ, Mueser KT. A meta-analysis of cognitive remediation in schizophrenia. Am J Psychiatry. 2007 Dec;164(12):1791-802. doi: 10.1176/appi.ajp.2007.07060906. PMID 18056233
- [Background] McMahon RP, Arndt S, Conley RR. More powerful two-sample tests for differences in repeated measures of adverse effects in psychiatric trials when only some patients may be at risk. Stat Med. 2005 Jan 15;24(1):11-21. doi: 10.1002/sim.1837. PMID 15515151
- [Background] Mozley LH, Gur RC, Gur RE, Mozley PD, Alavi A. Relationships between verbal memory performance and the cerebral distribution of fluorodeoxyglucose in patients with schizophrenia. Biol Psychiatry. 1996 Sep 15;40(6):443-51. doi: 10.1016/0006-3223(95)00421-1. PMID 8879463
- [Background] Nichols TE, Holmes AP. Nonparametric permutation tests for functional neuroimaging: a primer with examples. Hum Brain Mapp. 2002 Jan;15(1):1-25. doi: 10.1002/hbm.1058. PMID 11747097
- [Background] Nuechterlein KH, Barch DM, Gold JM, Goldberg TE, Green MF, Heaton RK. Identification of separable cognitive factors in schizophrenia. Schizophr Res. 2004 Dec 15;72(1):29-39. doi: 10.1016/j.schres.2004.09.007. PMID 15531405
- [Background] Park S, Holzman PS. Schizophrenics show spatial working memory deficits. Arch Gen Psychiatry. 1992 Dec;49(12):975-82. doi: 10.1001/archpsyc.1992.01820120063009. PMID 1449384
- [Background] Perrin F, Pernier J, Bertrand O, Echallier JF. Spherical splines for scalp potential and current density mapping. Electroencephalogr Clin Neurophysiol. 1989 Feb;72(2):184-7. doi: 10.1016/0013-4694(89)90180-6. PMID 2464490
- [Background] Ragland JD, Gur RC, Raz J, Schroeder L, Kohler CG, Smith RJ, Alavi A, Gur RE. Effect of schizophrenia on frontotemporal activity during word encoding and recognition: a PET cerebral blood flow study. Am J Psychiatry. 2001 Jul;158(7):1114-25. doi: 10.1176/appi.ajp.158.7.1114. PMID 11431234
- [Background] Saykin AJ, Gur RC, Gur RE, Mozley PD, Mozley LH, Resnick SM, Kester DB, Stafiniak P. Neuropsychological function in schizophrenia. Selective impairment in memory and learning. Arch Gen Psychiatry. 1991 Jul;48(7):618-24. doi: 10.1001/archpsyc.1991.01810310036007. PMID 2069492
- [Background] Weinberger DR, Egan MF, Bertolino A, Callicott JH, Mattay VS, Lipska BK, Berman KF, Goldberg TE. Prefrontal neurons and the genetics of schizophrenia. Biol Psychiatry. 2001 Dec 1;50(11):825-44. doi: 10.1016/s0006-3223(01)01252-5. PMID 11743939
- [Background] Wexler BE, Stevens AA, Bowers AA, Sernyak MJ, Goldman-Rakic PS. Word and tone working memory deficits in schizophrenia. Arch Gen Psychiatry. 1998 Dec;55(12):1093-6. doi: 10.1001/archpsyc.55.12.1093. PMID 9862552
- [Background] Wykes T, Brammer M, Mellers J, Bray P, Reeder C, Williams C, Corner J. Effects on the brain of a psychological treatment: cognitive remediation therapy: functional magnetic resonance imaging in schizophrenia. Br J Psychiatry. 2002 Aug;181:144-52. doi: 10.1017/s0007125000161872. PMID 12151286
- [Background] Westfall PH. 1997. Multiple testing of general contrasts using logical constraints and correlations, J Am Stat Assoc, 92; 299-306.
- [Background] Westfall PH, Tobias RD, Rom D, Wolfinger RD, Hochberg Y. Multiple comparisons and multiple tests using the SAS7 system, SAS Institute, Inc., Cary NC, pp. 149-175, 335-343, 1999.
- [Background] Schafer, JL. Analysis of Incomplete Multivariate Data, New York: Chapman and Hall. 1997
- [Background] Mattay VS, Goldberg TE, Fera F, Hariri AR, Tessitore A, Egan MF, Kolachana B, Callicott JH, Weinberger DR. Catechol O-methyltransferase val158-met genotype and individual variation in the brain response to amphetamine. Proc Natl Acad Sci U S A. 2003 May 13;100(10):6186-91. doi: 10.1073/pnas.0931309100. Epub 2003 Apr 25. PMID 12716966
- [Background] Little RJA, and Rubin DB. Statistical Analysis with Missing Data, Second Edition, New York: John Wiley & Sons, Inc. 2002.
- [Background] Cohen JD, Forman SD, Braver TS, Casey BJ, Servan-Schreiber D, Noll DC. Activation of the prefrontal cortex in a nonspatial working memory task with functional MRI. Hum Brain Mapp. 1994;1(4):293-304. doi: 10.1002/hbm.460010407. PMID 24591198
- [Background] Friedman D. ERPs during continuous recognition memory for words. Biol Psychol. 1990 Feb;30(1):61-87. doi: 10.1016/0301-0511(90)90091-a. PMID 2223937
- [Background] Holm S. A simple sequentially rejective multiple test procedure. Scandinavian Journal of Statistics, 6, 65-70, 1979.
- [Background] Kayser, J., Tenke, C.E. Consensus on PCA for ERP data, and sensibility of unrestricted solutions. Clinical Neurophysiology, 117(3), 703-707. (2006c).
- [Result] Kantrowitz JT, Sharif Z, Medalia A, Keefe RS, Harvey P, Bruder G, Barch DM, Choo T, Lee S, Lieberman JA. A Multicenter, Rater-Blinded, Randomized Controlled Study of Auditory Processing-Focused Cognitive Remediation Combined With Open-Label Lurasidone in Patients With Schizophrenia and Schizoaffective Disorder. J Clin Psychiatry. 2016 Jun;77(6):799-806. doi: 10.4088/JCP.15m09998. PMID 27035157
- [Derived] Roberts MT, Lloyd J, Valimaki M, Ho GW, Freemantle M, Bekefi AZ. Video games for people with schizophrenia. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD012844. doi: 10.1002/14651858.CD012844.pub2. PMID 33539561

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Remediation | Cognitive Activity Control Group
Started | 56 | 64
Completed | 33 | 41
Not Completed | 23 | 23

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Remediation | Cognitive Activity Control Group | Total
Number analyzed (Participants) | 56 | 64 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (9.9) | 38.1 (10.3) | 37.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 34 | 44 | 78

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Function Measured by MCCB Composite Score
Description: The MATRICS Consensus Cognitive Battery (MCCB) will be used to assess cognitive function. The MCCB composite score is comprised of sub-scale measures of: a) working memory; b) attention and vigilance; c) verbal learning; d) visual learning; e) speed of processing; f) reason and problem solving; and g) social cognition. The MCCB takes 90 minutes or less to complete.
  MCCB assessed 4 times: prestabilization (screening), randomization (after 6-8 weeks of lurasidone stabilization, prior to initial cognitive remediation), midpoint (after 20 cognitive remediation session), and study completion (final visit after 30 cognitive remediation sessions).
  MCCB composite scores are reported as t-scores where a t-score = 50 is the population average. Every 10 points is one standard deviation. There is no range as scores are as far from population average.
Time Frame: 4-6 month period
Population: Completers
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Remediation | Cognitive Activity Control Group
Number analyzed (Participants) | 33 | 41
units on a scale | 35.39 (11.99) | 30.73 (14.97)

2. Primary Outcome: Cognitive Function as Measured by the University of California, San Diego, Performance-Based Skills Assessment-Brief (UPSA-B) Scale
Description: The UPSA-B assesses functional capacity to perform tasks similar to those in daily life. Raw scores are converted into scaled scores ranging from 0-100, with higher scores indicating better functional capacity.
Time Frame: 4-6 month period
Population: Completed subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Remediation | Cognitive Activity Control Group
Number analyzed (Participants) | 33 | 40
units on a scale | 79.74 (10.99) | 75.85 (16.37)

3. Secondary Outcome: Cognition as Measured by Cognitive Assessment Interview (CAI)
Description: Cognitive Assessment Interview was used to obtain information about cognitive functioning from both subject and an informant. Composite CAI scores were reported. Scale ranges from 1-7 with the following anchors:
  1. Normal, no cognitive impairment
  2. Borderline impairment
  3. Mildly impaired
  4. Moderately impaired
  5. Markedly impaired
  6. Severely impaired
  7. Among the most extremely impaired
Time Frame: 4-6 month period
Population: completed subjects with available completed CAI data. Numbers above are correct as not all completed subjects (Analysis Population Description) had completed CAI assessment available for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Remediation | Cognitive Activity Control Group
Number analyzed (Participants) | 31 | 40
units on a scale | 2.74 (1.6) | 2.79 (1.18)

4. Secondary Outcome: Efficacy as Measured by Positive and Negative Syndrome Scale (PANSS)
Description: Total PANSS score with 30 items. Each item is rated 1-7 so the minimum Total PANSS score =30 and the maximum is 210. Anchors for each item are as follows, the higher values represent an increase in severity of symptoms:
  1. Absent
  2. Minimal
  3. Mild
  4. Moderate
  5. Moderately severe
  6. Severe
  7. Extremely severe
Time Frame: 4-6 month period
Population: Completed subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Remediation | Cognitive Activity Control Group
Number analyzed (Participants) | 33 | 41
units on a scale | 58.79 (14.71) | 61.1 (17.29)

ADVERSE EVENTS:
Arm/Group | Cognitive Remediation | Cognitive Activity Control Group
Serious Adverse Events (participants affected / at risk) | 5/56 | 7/64
Other Adverse Events (participants affected / at risk) | 0/56 | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Remediation (N=56) | Cognitive Activity Control Group (N=64)
Exacerbation (Nervous system disorders) | 4 (5) | 6 (7)
abnormal ECG (Cardiac disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes